CLINICAL TRIAL: NCT02383836
Title: Influence of Position on Detection of Patent Foramen Ovale by Simultaneous Transesophageal Echo and Transcranial Doppler
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0005-X14-HYMC
Record Dates: First submitted 2015-02-23; First posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Patent Foramen Ovale
Keywords: Patent Foramen Ovale
MeSH Terms: conditions — Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients will have simultaneous Transesophageal Echo (TEE) and Transcranial Doppler (TCD) performed and a comparison of timing, sensitivity and intensity of intravenously injected bubbles will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients needing a TEE evaluation to rule out a cardiac source of brain emboli

Exclusion Criteria:

* Patients unable to comply with protocol requirements
* Patients unable or unwilling to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a TEE with bubble injection to rule out a cardiac source of brain emboli following an acute neurological embolic event.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Bubble Detection | 3 minutes
  The amount of time until bubbles are detected will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel